CLINICAL TRIAL: NCT05797857
Title: Personalized Exercise Training to Improve Functional Capacity in Transthyretin Cardiac Amyloidosis
Brief Title: Exercise Training in Transthyretin Cardiac Amyloidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sarah Cuddy, MD, Cardiologist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022p002754
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Amyloid Cardiomyopathy; Transthyretin Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — A supervised, personalized exercise training program, which will consist of two 60-minute exercise training sessions per week.

SUMMARY:
Transthyretin cardiac amyloidosis causes debilitating heart failure in older adults. The proposed research will develop a personalized exercise training program to improve functional capacity in patients on optimal treatment for transthyretin cardiac amyloidosis. This is a vital next step to improve functional capacity and quality of life of people suffering from transthyretin cardiac amyloidosis.

DETAILED DESCRIPTION:
Heart failure (HF) affects over 5 million adults over the age of 65. Cardiac transthyretin amyloidosis (ATTR-CM) is a cause of HF in ~10% of older adults and leads to significant morbidity and mortality. Exercise intolerance is traditionally attributed to cardiac dysfunction but the contribution of other systems to this has not been studied. Musculoskeletal involvement is common in ATTR-CM and occur 5-10 years prior to onset of HF. Tafamidis, a transthyretin stabilizer, is the only approved treatment for ATTR-CM. It slows disease progression, prolongs life, and reduces HF hospitalizations. However, it does not improve functional capacity- no therapeutic intervention has been shown to do so in ATTR-CM.

The idea behind this project is that skeletal muscle dysfunction from amyloidosis and HF severely limits exercise capacity and, thus, quality of life in ATTR-CM, and that targeted exercise training will improve quality of life by improving skeletal muscle performance and aerobic capacity. Cardiopulmonary exercise testing (CPET) and the short physical performance battery (SBBP), including a leg extensor muscle power assessment will be used to achieve the following specific aims; 1) to compare skeletal muscle performance in ATTR-CM and non-amyloid HF; and 2) to determine improvements in aerobic capacity and quality of life due to 12 weeks of supervised exercise training in patients with ATTR-CM. To achieve the second aim, we will use a personalized exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis and typing of ATTR-CM by endomyocardial biopsy or by Grade 2 or Grade 3 pyrophosphate (PYP) positivity (exception: nonamyloid control arm in aim 1).

  * Diagnosis of heart failure, with prior or current need of diuretics and increased N-terminal prohormone B-natureitic peptide (BNP) (≥450 pg/ml).
  * Peak VO2 <80% predicted, indicating impaired aerobic capacity (for aim 2 only).
  * Taking tafamidis (for aim 2 only)
  * Able to walk 4 meters (with or without the use of an assistive device) and independent with basic activities of daily living at the time of enrolment.
  * Adequate clinical stability has been achieved in the judgment of the investigator to allow participation in study assessments and the intervention.
  * Signed informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

* Acute myocardial infarction (Note: given that cardiac biomarkers such as troponin are frequently elevated in ATTR-CM patients, the diagnosis of acute myocardial infarction should be based on clinical diagnosis, not biomarkers alone)

  * >70% obstructive coronary artery disease
  * Severe aortic valve stenosis
  * Already actively participating in formal, facility-based cardiac exercise
  * Already engaging in regular moderate to vigorous exercise conditioning defined as > 30 minutes per day, ≥ twice per week consistently during the previous 6 weeks
  * Ventricular assist device
  * Light chain amyloidosis or other form of non-ATTR amyloidosis
  * Advanced chronic kidney disease defined as estimated glomerular filtration rate <20 mL/min/1.73m2
  * Any organ transplantation
  * Terminal illness other than HF with life expectancy < 1 year
  * Pacemaker or implantable cardioverter-defibrillato (ICD) with heart rate limits < expected heart rates for exercise and unable to be reprogrammed
  * Neuropathy due to transthyretin (TTR) mutation
  * Impairment from stroke, injury or other medical disorder that precludes participation in the intervention
  * Abnormal cardiopulmonary exercise testing (CPET) finding that requires further investigation and management
  * Dementia that precludes ability to participate in exercise and follow study protocols
  * High risk for non-adherence as determined by screening evaluation
  * Inability or unwillingness to comply with the study requirements

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
peak oxygen consumption (VO2) | 12 weeks
  CPET performed at baseline and 12-weeks, following the exercise intervention will be used to measure aerobic capacity, peak VO2. The change in peak VO2 from baseline to 12 weeks is the primary outcome measure. An increase of > 1.0 ml/kg/min is considered a clinically meaningful increase

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire | 12 weeks
  Kansas City Cardiomyopathy Questionnaire (KCCQ) is a quality of life questionnaire. This will be recorded at baseline, 4-weeks and 12-weeks. The change in KCCQ score from baseline to 12 weeks is a secondary outcome. KCCQ scores are scaled from 0 to 100; where 0 denotes the lowest reportable health status and 100 the highest. An increase of 5 points is considered a clinically meaningful increase.
Lower extremity function | 12 weeks
  The short physical performance battery (SPPB) is an assessment of lower extremity function. The change in SPPB score from baseline to 12 weeks is a secondary outcome. This is a scale of 0-12, where 0 denotes the worst performance and 12 the highest. An increase of 1 point is considered a clinically meaningful increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
A limited access dataset generated from this project will rapidly be made available to the broader community for distribution to outside researchers according to established Mass General Brigham and NHLBI procedures and in accordance with NIH policies. Exercise training plans developed as part of this proposal will be made available.